CLINICAL TRIAL: NCT01120132
Title: A Multi-Center, Randomized, Double-Masked Evaluation of the Efficacy of Administration of FOV1101-00 (Cyclosporine Low Dose and High Dose) and Prednisolone Acetate Compared to Its Components and Vehicle in Patients With Mild Ongoing Ocular Allergic Inflammation
Brief Title: Study Evaluating the Efficacy of Administration of Cyclosporine (Low Dose and High Dose) and Prednisolone Acetate Compared to Its Components and Vehicle in Patients With Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fovea Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FOV1101/CLIN202; 10-003-03 (Other: ORA Inc)
Record Dates: First submitted 2010-04-29; First posted 2010-05-10 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cyclosporine low dose , Prednisolone Acetate (Experimental): Administration of a solution of Cyclosporine (low dose) and a suspension of Prednisolone Acetate
  Interventions: Drug: CsA low dose; Drug: PA
- Cyclosporine high dose, Prednisolone Acetate (Experimental): Administration of a solution of Cyclosporine (high dose) and a suspension of Prednisolone Acetate
  Interventions: Drug: CsA high dose; Drug: PA
- Cyclosporine high dose (Experimental): Administration of a solution of Cyclosporine (high dose) and Placebo
  Interventions: Drug: CsA high dose; Drug: Placebo
- Cyclosporine low dose (Experimental): Administration of a solution of Cyclosporine (low dose) and Placebo
  Interventions: Drug: CsA low dose; Drug: Placebo
- Prednisolone Acetate (Active Comparator): Administration of a suspension of Prednisolone Acetate and Placebo
  Interventions: Drug: PA
- Placebo (Placebo Comparator): Administration of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CsA high dose — Solution of Cyclosporine (high dose) administered during 28 days
  Arms: Cyclosporine high dose; Cyclosporine high dose, Prednisolone Acetate
Drug: CsA low dose — Solution of Cyclosporine (low dose) administered during 28 days
  Arms: Cyclosporine low dose; Cyclosporine low dose , Prednisolone Acetate
Drug: PA — Suspension of Prednisolone Acetate administered during 28 days
  Arms: Cyclosporine high dose, Prednisolone Acetate; Cyclosporine low dose , Prednisolone Acetate; Prednisolone Acetate
Drug: Placebo — Placebo solution administered during 28 days
  Arms: Cyclosporine high dose; Cyclosporine low dose; Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of the administration of cyclosporine and prednisolone acetate compared to placebo in the treatment of allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* history of ocular allergies and a positive skin test reaction to perennial allergens within the past 24 months and a history of chronic eye irritation
* visual acuity score ≥ 0.60 (EDTS)
* negative urine pregnancy test for female patients, and use of adequate birth control throughout the study period.

Exclusion Criteria:

* active ocular infection; preauricular lymphadenopathy or ocular condition that could affect study; glaucoma or abnormal intraocular pressure; ocular surgery within past 3 months; history of asthma, pregnancy or nursing
* contraindications or known allergies to the study drug(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Diary assessment of signs and symptoms of ocular allergy | During the 28 days of treatment
  Patient-reported ocular itching and redness

SECONDARY OUTCOMES:
Diary and office assessments of various ocular and nasal allergy signs and symptoms | During 28 days of treatment
  Patient-reported ocular itching and redness, lid swelling, tearing and nasal itching
  Investigator assessments of ocular redness and chemosis
Safety | During the 28 days of treatment
  Ocular tolerance and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Louise Jacques, MD MBA, Study Chair — Fovea Pharmaceuticals SA
Locations (1):
- ORA, Andover, Massachusetts, United States